# **Informed Consent Form**

Official Title: Messages About Reduced Nicotine in Combusted Tobacco Products

NCT Number: NCT05506046

**Document Date:** 06/06/2022

## Georgia State University School of Public Health Informed Consent

Title: Communicating about Nicotine and Differential Risks of Tobacco Products

Principal Investigator: Lucy Popova, PhD Sponsor: National Institutes of Health

## I. Purpose:

The purpose of the study is to learn about how best to communicate about harms of nicotine and different tobacco products. You are invited to take part because you are an adult above the age of 18. A total of 1,800 people will be recruited for this study. This study involves two parts, including a 15-minute survey now and a 5-minute survey in two weeks.

#### II. Procedures:

You are being asked to take part in a research study. If you decide to participate, you will take two online surveys. The first survey will take about 15 minutes of your time. You will see some messages about various topics and products you may be familiar with. You will be asked to evaluate these messages and what you think and how you feel after seeing the messages. You will also answer questions about your tobacco use and views.

#### III. Risks:

In this study, you will not have any more risks than you would in a normal day of life.

### IV. Benefits:

Your answers will help us understand how people think and feel about several consumer products. The results of this study will help future research.

#### V. Compensation:

You will receive points based on your existing agreement with Ipsos/KnowledgePanel for participating in this study.

## VI. Voluntary Participation and Withdrawal:

Participation in research is voluntary. You do not have to be in this study. If you decide to be in the study and change your mind, you have the right to drop out at any time. You can skip questions or stop at any time. Whatever you decide, you will not lose any benefits you would have had otherwise.

## VII. Confidentiality:

Version Date: 6/6/2022

We will keep your records private to the extent allowed by law. Dr. Popova and GSU research staff will have access to the information you give. Information may also be shared with those who make sure the study is done correctly (GSU Institutional Review Board, the Office for Human Research Protection (OHRP), and the National Institutes of Health). We will use an ID number rather than your name on study records. The GSU researchers will not have access to your personal information. The survey answers you provide will be stored in a secured database that does not have personal information. Your name and other facts that might point to you will not appear when we present this study or publish its results. The findings will be summarized and reported in group form. You will not be identified personally.

#### VIII. Contact Persons:

Contact Dr. Lucy Popova at 404-413-9338 or via email at lpopova1@gsu.edu if you have questions, concerns, or complaints about this study. You can also call if you think you have been harmed by the study.

Contact the GSU Office of Human Research Protections at 404-413-3500 or irb@gsu.edu

- if you have questions about your rights as a research participant
- if you have questions, concerns, or complaints about the research

#### IX. Clinical trial information:

A description of this clinical trial will be available on https://clinicaltrials.gov/, as required by U.S. Law. This Web site will not include information that can identify you. At most, the Web site will include a summary of the results. You can search this Web site at any time.

X. Copy of Consent Form to Participant:

You may print a copy of the consent form for your records.

If you want to volunteer for this research, please click continue.

Version Date: 6/6/2022